CLINICAL TRIAL: NCT00165022
Title: Development of a Novel Disease-Specific Quality of Life Questionnaire for Gastroesophageal Reflux Disease (GERD) Patients in Chinese Population
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Other Study IDs: GQOL
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
A questionnaire composed of items addressing psychological, emotional and social aspects of GERD is developed for Chinese population. We plan to conduct a validation study on this novel disease-specific quality of life (QoL) instrument. This study aims to evaluate various indicators of validity and reliability, which include criterion validity, test-retest reliability, responsiveness, internal consistency reliability and discriminant validity.

After initial pilot testing of face validity and content validity, two hundred GERD patients from the gastroenterology and ulcer clinics of cluster NTE hospitals will be invited to complete a revised 18-item version of GERD-QOL questionnaire. The data from GERD QOL will be evaluated using exploratory factor analysis to identify appropriate items and domains and the internal consistency of the domains will be determined and further refinement of questionnaire will follow.

100 GERD patients will complete GERD-QOL, SF-36 health survey and the visual analog scale (VAS) questionnaire for criterion validation. 100 GERD patients with stable symptom profile will repeat GERD QOL two weeks after the first administration for evaluation of test-retest reliability.

Another 26 patients who are receiving maintenance acid suppressive therapy and in remission of symptom will be recruited as controls for comparison with active reflux patients. The ability to distinguish active patients from controls in remission is known as discriminant validity.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with 1 attack of heartburn and/or acid regurgitation per week as chief complaint in recent 6 months

Exclusion Criteria:Patients with

* GERD as GI involvement of systemic disease e.g. scleroderma, SLE, thyrotoxicosis, chronic intestinal pseudo-obstruction
* Cause of esophagitis other than GERD e.g. drug induced, infection, nasogastric tube injury
* Previous gastrointestinal or hepatobiliary surgery (including cholecystectomy)
* Organic pathology of upper GI tract that may present as reflux / dyspeptic symptom e.g. peptic ulcer, gastric cancer, gastric outlet obstruction
* Presence of alarm symptom that does not suggest functional GI disorder
* Use of NSAID in recent 4 weeks (Low dose aspirin < 300 mg is allowed)
* Pregnant woman or lactating female
* Illiterate patient (who cannot administer questionnaire)
* Known hypersensitivity to PPI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2003-09; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin CY WU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, China